CLINICAL TRIAL: NCT04309162
Title: Soft Tissue Therapy in Managing Procedural Pain Among Neonates Admitted in Neonatal Intensive Care Unit: A Single Group, Pretest Posttest Quasi Experimental Study.
Brief Title: Soft Tissue Therapy in Managing Procedural Pain Among Neonates.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asir John Samuel (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Associate Professor Maharishi Markandeshwar (Deemed to be university), Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMDU/IEC/1528; U1111-1249-2317 (Other: Universal Trial Number (UTN) by WHO ICTRP)
Record Dates: First submitted 2020-03-06; First posted 2020-03-16 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Neonatal Disorder
Keywords: Neonatal; Newborns; Infant; NICU; Procedural Pain; Massage Therapy
MeSH Terms: conditions — Infant, Newborn, Diseases; Pain, Procedural | interventions — Therapy, Soft Tissue

STUDY DESIGN:
Intervention Model Description: A single group Pretest-Posttest quasi experimental design
Masking Description: The neonates admitted in NICU are masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- soft tissue therapy (Experimental): Soft tissue therapy includes various techniques which is usually done by manipulating the soft tissues. The techques like stroking, petrissage, percussing maniulations are proved helpful in managing various painful conditions. The main effect of the soft tissue therapy is enhanced blood circulation to the area. When the techniques of soft tissue therapy are applied they will results in stretching and rubbing the muscular tissue which results in increased venous flow to heart and removal of the lactic acid accumulation occurs as the fresh supply of blood to the area will increased. Endorphins the natural pain relievers are released as there is improved oxygenation and perfusion of oxygen in tissues.
  Interventions: Other: Soft tissue therapy

INTERVENTIONS:
Other: Soft tissue therapy — Soft tissue therapy consists of various soft tissue manipulating techniques which includes the stroking, percussive and tapping manipulations. The treatment techniques are divided according to the body parts. under this techniques are tapping, flat finger kneading, Stroking, skin rolling etc.

SUMMARY:
Effect of Soft tissue Therapy in managing Procedural Pain among neonates admitted in neonatal intensive care unit. This study focuses on the Procedural pain management with the help of Soft tissue manipulation which includes various techniques like stroking, petrissage manipulations.

DETAILED DESCRIPTION:
Background: Neonatal intensive care unit (NICU) is a specialized unit created for sick and premature newborns. There are various painful procedures through which neonates have to undergo during the NICU stay. The most common procedure is the blood tests for the laboratory investigations which include the heel lancing and venipuncture. Pain is the one of the cause of the development of the acute stress in neonates soft tissue therapy has considered as the major contributory factor of in reducing the procedural pain among neonates admitted NICU. There is no documentation on soft tissue therapy in managing procedural pain in neonates.

Purpose: To determine the effects of soft tissue therapy in managing procedural pain among neonates admitted in NICU.

Methods and materials: The study will recruit neonates who underwent for various painful procedures in NICU such as venous and arterial puncture, capillary puncture, pulmonary mechanical ventilation, tracheal intubation, removal of adhesive tapes, the introduction of various drains etc. Preterm, Term, Full terms Neonates Stable Neonates. The samples will be taken via stratified random sampling technique. Neonates with unstable vitals are to be excluded from the study.

Discussion: To best of our knowledge, this will be the first study determining the effects of soft tissue therapy in procedural pain on neonates admitted in NICU. The role of neonatal physiotherapist in NICU is to provide diagnosis and treatment to admitted newborns. Massage therapy is considered as an effective management technique in pain management. In this study soft tissue therapy will be applied to neonates especially in context with procedural pain. There are various painful procedures performed to check the prognosis of neonates.

Keywords: Neonatal; Newborns; Infant; NICU; Procedural pain; Massage therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates who underwent various painful procedures in NICU such as venous, arterial and capillary puncture, mechanical ventilation for pulmonary causes, tracheal intubation, adhesive tapes removal, insertion of various drains etc.
2. Preterm, Term, Post terms Neonates
3. Stable Neonates.

Exclusion Criteria:

1. Post-Surgical cases
2. Parents of Neonates who are not willing to enroll their infant in study.
3. Neonates with congenital anomalies.
4. Neonates with extreme low birth weight.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Neonatal Infant Pain Scale (NIPS) | Baseline, 4 days after the intervention.
  Neonatal Infant Pain Scale is basically a behavioral tool and can be used in preterm and full term infants. The total score is 7. NIPS score is divided into 3 categories. 0-2 indicates no pain, 3-4 mild to moderate pain, >4 indicates severe pain.

SECONDARY OUTCOMES:
Change in Neonatal Pain Agitation and sedation scale(N-PASS) | Baseline, 4 days after the intervention
  N-PASS is scale which is used to assess Procedural, postoperative mechanically . ventilated patients. It includes variables like crying, irritability, facial expression, extremity tone and vital signs. It is 0 to 10 scale high level of score indicates more aggression and intense behavior and low levels indicates decreased level of stimulation and deeper sedation.

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Sharma, BPT, Principal Investigator — Maharishi Markandeshwar institute of Physiotherapy and Rehabilitation; Asir J Samuel, MPT, PhD, Study Chair — Maharishi Markandeshwar institute of Physiotherapy and Rehabilitation; Neha Sharma, MPT, Study Director — Maharishi Markandeshwar institute of Physiotherapy and Rehabilitation
Locations (1):
- Abhishek Sharma, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brummelte S, Grunau RE, Chau V, Poskitt KJ, Brant R, Vinall J, Gover A, Synnes AR, Miller SP. Procedural pain and brain development in premature newborns. Ann Neurol. 2012 Mar;71(3):385-96. doi: 10.1002/ana.22267. Epub 2012 Feb 28. PMID 22374882
- [Result] Niemi AK. Review of Randomized Controlled Trials of Massage in Preterm Infants. Children (Basel). 2017 Apr 3;4(4):21. doi: 10.3390/children4040021. PMID 28368368
- [Result] Field T, Diego M, Hernandez-Reif M. Preterm infant massage therapy research: a review. Infant Behav Dev. 2010 Apr;33(2):115-24. doi: 10.1016/j.infbeh.2009.12.004. PMID 20137814
- [Result] Jain S, Kumar P, McMillan DD. Prior leg massage decreases pain responses to heel stick in preterm babies. J Paediatr Child Health. 2006 Sep;42(9):505-8. doi: 10.1111/j.1440-1754.2006.00912.x. PMID 16925535
- See also: Preterm infants are exposed to various painful procedures in Neonatal intensive care unit. Early Procedural pain exposure results int the harmful effects on the development of brain. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3760843/
- See also: randomized controlled trials on the effects of massage in preterm infants suggest improved weight gain and shortened length of hospital stay. Improved weight gain may be mediated through increase in vagal tone but more studies are needed. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2844909/
- See also: Massage therapy is considered as the effective non pharmacological measure for reducing the procedural pain in NICU and reduces their hospital stay. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5406680/
- See also: By applying massage therapy before doing heel stick procedure pain responses are reduced in preterm infants — https://www.ncbi.nlm.nih.gov/pubmed/16925535/